CLINICAL TRIAL: NCT05150600
Title: Inverse Ratio Ventilation Versus Conventional Ratio Ventilation During One Lung Ventilation in Neonatal Open Repair of Esophageal Atresia/Tracheoesophageal Fistula: A Randomized Clinical Trial.
Brief Title: Inverse Ratio Ventilation in Neonatal Open Repair of Tracheoesophageal Fistula.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Akram Mohamed Mohamed Amer, Lecturer in the department of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R172/2021
Record Dates: First submitted 2021-11-12; First posted 2021-12-09 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Tracheo Esophageal Fistula
Keywords: Inverse ratio Ventilation; Neonates; Esophageal atresia/Tracheoesophageal fistula; one lung ventilation
MeSH Terms: conditions — Tracheoesophageal Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Inverse Ratio Ventilation (IRV) (Experimental): The inspiratory to expiratory (I:E) ratio in this group will be 2:1 with the maximum inspiratory time (Ti) of 1.3 seconds
  Interventions: Procedure: Inverse Ratio Ventilation
- Group Conventional Ratio Ventilation (CRV) (No Intervention): The inspiratory to expiratory (I:E) ratio in this group will be 1:2 with the minimum inspiratory time (Ti) of 0.4 seconds

INTERVENTIONS:
Procedure: Inverse Ratio Ventilation — The inspiratory to expiratory (I:E) ratio will be reversed to be 2:1 during mechanical ventilation
  Arms: Group Inverse Ratio Ventilation (IRV)

SUMMARY:
Background and Objectives: Maintaining oxygenation during neonatal open repair of esophageal atresia is difficult. Inverse ratio ventilation can be used during one lung ventilation (OLV) to improve the oxygenation and lung mechanics. The investigators will compare inverse ratio to conventional ratio ventilation during OLV in neonatal open repair of esophageal atresia regarding effect in oxygenation, hemodynamic variables, incidence of complications, and easiness of procedure.

Methods: The investigators will enroll 40 term neonates undergoing open right thoracotomy for esophageal atresia repair in this prospective randomized study. The patients will be randomly assigned into 2 groups based on inspiratory to expiratory (I:E) ratio of mechanical ventilation parameters (I:E ratio will be 2:1 in IRV and 1:2 in CRV). The incidence of desaturation episodes that needs to stop the procedure and reinflation of the lung will recorded as the primary outcome while hemodynamic parameters, incidence of complications, and length of surgical procedure will be recorded as the secondary outcomes.

DETAILED DESCRIPTION:
INTRODUCTION:

Maintaining adequate oxygenation after lung retraction and one lung ventilation (OLV) in open thoracotomy during neonatal repair of esophageal atresia/ tracheoesophageal fistula is extremely difficult and usually required stopping the procedure and reinflation of the retracted lung which prolong the surgery time, stopping the procedure during critical situations and endanger the fragile neonate from hypoxemia.

Inverse ratio ventilation has been used originally for long time in patients with acute respiratory distress syndrome (ARDS) to improve the oxygenation and lung function. The mechanism with inverse ratio ventilation is to prolong the inspiratory time with reducing the airway pressure and elevate the mean airway pressure preventing the alveoli from collapse. Also inverse ratio ventilation (IRV) used in many studies in adults during OLV with better oxygenation and lung mechanics.

Despite the standard ventilatory sitting in neonatal anesthesia is to adjust the inspiratory time to achieve inspiratory to expiratory (I:E) ratio of 1:2 to 1:3, but inverse I:E ratio (with inspiratory time longer than expiratory time) up to 4:1 in neonatal mechanical ventilation has been shown to be effective in improving oxygenation, PaO2, and gas distribution in atelectatic lungs. Inverse I:E ratio in neonatal mechanical ventilation should be used in caution and for a short period of time to avoid possible complications as air trapping/auto PEEP, volutrauma, air leaks, decrease venous return, and increase pulmonary vascular resistance.

AIM/ OBJECTIVES:

1. To compare the incidence of desaturation episodes that needs to stop the procedure and reinflation of the lung using inverse ratio ventilation versus conventional ratio ventilation during one lung ventilation in neonatal open repair of esophageal atresia/tracheoesophageal fistula.
2. To determine the effect of inverse ratio ventilation on hemodynamic parameters, incidence of complications, and length of surgical procedure as compared to conventional ratio ventilation.

METHODOLOGY:

The study will be conducted at Ain Shams University Hospitals after ethical committee approval and obtaining an informed written consent from patients' parents or legal guardian.

* Type of Study Prospective randomized controlled clinical trial.
* Study Setting Pediatric surgery operating theatre in Ain shams university hospital, Cairo, Egypt.
* Study Period The study will be started immediately after ethical committee approval starting from October 2021 aiming to be completed within 6 months.
* Study Population

  * Inclusion Criteria: The patients will be of ASA physical status II-III, neonates aged less than 28 days and undergoing open repair of esophageal atresia/ tracheoesophageal fistula with right thoracotomy. All patients' will be full term with gestational age ≥ 36 weeks and weigh ≥ 2.5 kilograms.
  * Exclusion Criteria: Significant congenital heart disease including cyanotic heart disease, single ventricle pathology, large intracardiac defect with significant left to right shunt, and severe pulmonary hypertension more than 50 mmHg. Other exclusion criteria included prematurity, pneumonia or severe chest infection prior to the surgery, and parent or guardian refusal.
* Sampling Method Based on inspiratory to expiratory (I:E) ratio used in positive pressure ventilation, patients will be randomly and evenly assigned to one of two groups (20 patients each) using a computer-generated list: experimental group IRV (inverse ratio ventilation) and control group CRV (conventional ratio ventilation).

Group IRV: the I:E ratio in this group will be 2:1 with the maximum inspiratory time (Ti) of 1.3 seconds.

Group CRV: the I:E ratio in this group will be 1:2 with the minimum inspiratory time (Ti) of 0.4 seconds.

* Sample Size Sample size was calculated using PASS 11.0 and based on a study carried out by Son et al., 2020. Group sample size of 20 patients in Group one and 20 patients in Group two achieve 82% power to detect a difference between the group proportions of 0.4000. The proportion in group one (the treatment group) is assumed to be 0.1000 under null hypothesis and 0.5000 under the alternative hypothesis. The proportion in group two (the control group) is 0.1000. The test statistic used is the two-sided Z test with pooled variance. The significance level of the test was targeted at 0.0500. The significance level actually achieved by this design is 0.0361. The sample size was inflated by 10% to account for attrition problem in prospective studies.
* Ethical Considerations After acquiring local medical ethics committee approval and informed written consent from the parent or guardian, The investigators will enroll 40 patients in this study.
* Study Tools AND/ OR Study Procedures AND/OR Study Interventions All included patients will be admitted to neonatal intensive care unit (NICU) and kept Nil Per Os (NPO) after establishing the diagnosis of esophageal atresia/tracheoesophageal fistula, had a secured venous access and received dextrose containing intravenous fluid according to the orders given by the neonatologist. An umbilical artery catheter will be inserted by the neonatologist prior to the surgery, also an orogastric tube (OGT) will be inserted in the proximal esophageal pouch and a low negative pressure suction will be applied to suck any secretions in the esophagus and decrease risk of aspiration.

Another intravenous (iv) cannula will be inserted after induction of anesthesia and a femoral 22 gauge (G) arterial line will be inserted in any patient without an umbilical artery catheter.

After applying standard monitors (non-invasive blood pressure, 5-lead ECG and 2 pulse oximetry; one pre-ductal and one post-ductal, 2 temperature probes; one oropharyngeal and one axillary), anesthesia induction will be started with inhalational anesthetics sevoflurane 2% in 100% oxygen and increasing gradually till end-tidal sevoflurane reach 4-6% with maintaining spontaneous breathing to avoid gastric distension with positive pressure ventilation (PPV) then tracheal intubation will be facilitated with lidocaine 10% topical spray one puff applied to the glottic opening just before insertion of 3 or 3.5 mm non-cuffed endotracheal tube (ETT), then ETT will be fixed just above the tracheal carina (confirmed by auscultation -the ETT will be initially pushed endobronchial then gradually withdrawn till bilateral breath sound heard- and absence of gastric distension with gentle positive pressure ventilation).

After ensure the correct position of ETT just above the carina and below the tracheoesophageal fistula and the patient hemodynamically stable, positive pressure ventilation will be started after establishing muscle relaxation with atracurium 0.5 mg/kg. Anesthesia will be maintained with sevoflurane 1-2% in oxygen/air mixture and fentanyl infusion of 1-2 mcg/kg/h. Fraction of inspired oxygen (FiO2) will be maintained to the lower limit to keep oxygen saturation (SpO2) ≥ 92% with minimum FiO2 of 0.3. IV fluids will be maintained as preoperative rate with boluses of normal saline will be given to replace blood loss and third space loss. Blood transfusion will be given in cases lost more than 10% of their total blood volume.

All patient will be mechanically ventilated with synchronized intermittent mandatory ventilation-pressure controlled ventilation (SIMV-PCV) mode with the following parameters; peak inspiratory pressure (PIP) 10-15 cmH2O above positive end-expiratory pressure (PEEP) of 5 cmH2O to achieve expired tidal volume (VTE) from 7-10 ml/kg, Respiratory rate (RR) ranging from 30 to 50 breath/minute to achieve end-tidal CO2 (EtCO2) from 30 mmHg up to 50 mmHg, and pressure support (PS) 12 cmH2O.

The same pediatric surgery team will perform all procedures. After positioning of the patient in the right lateral position, the right hemithorax will be opened then the right lung will be retracted to expose and ligate the fistula then end to end esophageal anastomosis will be performed. The right lung will be re-inflated under direct vision to ensure full lung expansion after finishing of esophageal anastomosis then the right hemithorax will be closed with chest tube in situ. Patients in IRV group will resumed conventional I:E ratio ventilation after resuming two lungs ventilation.

Hemodynamic variables including heart rate (HR), mean arterial pressure (MAP), and oxygen saturation (SpO2) will be recorded: baseline (before induction of anesthesia), before initiation of PPV, after the initiation of PPV, after initiation of OLV and every 10 min until the end of the procedure.

The incidence of hypotension (as the lower limit of normal mean BP on the day of birth, in mmHg, is approximately equal to the gestational age in weeks, so hypotension considered if MAP is less than the gestational age in weeks); and bradycardia (defined as: HR< 90 beats/min, as the lower limit of normal HR in sleeping neonate is 90 beats/min) or hypoxemia (oxygen saturation less than 90%) will be recorded.

In cases of hypotension, the patient will be treated initially with an IV fluid bolus of 10-20 ml/kg normal saline over 5-10 minutes. In case of estimated blood loss exceeded 10% of TBV, transfusion of packed red blood cells (PRBCs) of 10-15 ml ml/kg over 10-20 minutes will be given. If the hypotension persisted despite of volume loading, dopamine IV infusion will be used in dose range 5-10 mcg/kg/min until the blood pressure normalize. Bradycardia will be treated initially with stopping the surgery and manual reinflation of right lung if associated with hypoxia and if persisted or not related to hypoxia will be treated with intravenous atropine 0.02 mg/kg.

In the case of a drop in oxygen saturation of less than 90%, the FiO2 and the PEEP will be increased to 1 and 7 cmH2O respectively, and if desaturation persist, the surgery will be stopped with manual reinflation of right lung.

The incidence of stopping the procedure for manual reinflation of the lung will be recorded, also the length of the surgical procedure starting from skin incision till skin closure will be recorded.

Arterial blood gases (ABG) sample will be done two times during the procedure; first one after established positive pressure ventilation by 10 minutes and before the surgical incision, the second sample will be done after established OLV by 10 minutes but not during desaturation episode. SaO2, PO2 and PCO2, will be recorded.

After completion of the procedure, patients will be transferred to the NICU intubated, ventilated and sedated. In the NICU chest X-ray will be performed immediately after patient arrival to exclude pneumothorax.

The incidence of complications including desaturation episodes that needs only increase FiO2 and/or PEEP, desaturation episodes that needs stop the procedure with lung reinflation, hypotension, bradycardia, hypercapnia, needs for vasopressor and blood loss exceeding 10% from TBV will be recorded.

Intraoperative and postoperative data will be collected by the an anesthesia resident not participating in the study.

* Statistical Analysis Numerical data are presented as the mean (standard deviation) or median (range) while categorical data are presented as the number of cases (percentage). Between-group comparisons of numerical variables will be performed by the independent sample T-test, or Mann-Whitney test as appropriate, while those of categorical variables will be performed by the Chi-square test. For all tests, a P (probability) value < 0.05 will be considered statistically significant.
* Statistical Package The data collected will be analyzed with statistical program SPSS (version 22.0 Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* The patients will be of ASA physical status II-III, neonates aged less than 28 days and undergoing open repair of esophageal atresia/tracheoesophageal fistula with right thoracotomy. All patients' will be full term with gestational age ≥ 36 weeks and weigh ≥ 2.5 kilograms.

Exclusion Criteria:

* Significant congenital heart disease including cyanotic heart disease, single ventricle pathology, large intracardiac defect with significant left to right shunt, and severe pulmonary hypertension more than 50 mmHg. Other exclusion criteria included prematurity, pneumonia or severe chest infection prior to the surgery, and parent or guardian refusal.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of severe desaturation episodes | 6 months
  Incidence of desaturation episodes that needs to stop the procedure and reinflation of the retracted lung.

SECONDARY OUTCOMES:
Mean blood pressure | 6 months
  We will test the effect of inverse ratio ventilation in mean blood pressure measured in millimeter mercury "mmHg" compared to conventional ratio ventilation.
Incidence of complications | 6 months
  We will test the effect of inverse ratio ventilation in incidence of complications (including hypotension, bradycardia, desaturation, and pneumothorax "measured as a percentage") compared to conventional ratio ventilation.
Length of surgical procedure | 6 months
  We will test the effect of inverse ratio ventilation on length of surgical procedure (measured in minutes) compared to conventional ratio ventilation.
Heart rate | 6 months
  We will test the effect of inverse ratio ventilation in heart rate measured in beats per minutes compared to conventional ratio ventilation.
Oxygen saturation | 6 months
  We will test the effect of inverse ratio ventilation in oxygen saturation measured in percentage compared to conventional ratio ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Akram Amer, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams university- faculty of medicine- department of anesthesia, intensive care and pain management, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through the study may be provided to qualified researchers with academic interest in neonatal anesthesia. Data shared will be coded, with no patient health information included.
Supporting Information: Study Protocol, CSR
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. For more information or to submit a request, please contact akram.amer@med.asu.edu.eg